CLINICAL TRIAL: NCT01998308
Title: Intra-articular Hyaluronic Acid Knee Injection: Randomized Control Trial.
Brief Title: Comparison Between Four Types of Single Dose Hyaluronic Acid Injection in Patients With Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Mahmoud A Hafez, MSc Orth, Dip SICOT, FRCS Ed, MD, Mahmoud A Hafez, October 6 University
Other Study IDs: October6U-0001
Record Dates: First submitted 2013-11-16; First posted 2013-11-28 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Gels; Hyaluronic Acid

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: 50 Knees will have single injection of Crespine gel
  Interventions: Drug: Crespine gel
- Group 2: 50 Knees will have single injection of 2 ampules of intragel
  Interventions: Drug: Intragel
- Group 3: 50 knees will have single injection of crespine plus gel
  Interventions: Drug: Crespine plus gel
- Group 4: 50 knees will have single injection of Monovisc
  Interventions: Drug: Monovisc

INTERVENTIONS:
Drug: Crespine gel — 50 Knees will have single injection of Crespine gel
  Groups: Group 1
Drug: Intragel — 50 Knees will have single injection of 2 ampules of Intragel
  Groups: Group 2
Drug: Crespine plus gel — 50 Knees will have single injection of Crespine Plus Gel
  Groups: Group 3
Drug: Monovisc — 50 Knees will have single injection of Monovisc
  Groups: Group 4

SUMMARY:
Study design:

Allocation: Randomized. Endpoint Classification: Comparative Study. Intervention model: Parallel Assignment. Masking: Double Blind (Subject, Assessed) Primary purpose: Comparison.

Official Title: Intra-articular hyaluronic acid knee injection: randomized control trail.

Primary outcome measures:

* Lower extremity functional scale
* Visual analogue scale
* Range of motion
* Kellgren and Lawrence class grade Estimated enrollment: 100 Study start date: December 2012 Estimated study completion date: June 2013 Estimated primary completion date: December 2013

DETAILED DESCRIPTION:
The study include:

200 knees, 50 knees will have single injection of Crespine gel, and 50 knees will have single injection of 2 ampules of Intragel, also 50 knees will have single injection of Crespine plus gel and 50 knees will have single injection of Monovisc The patient will be randomized to Crespine gel or to Intragel, and Crespine Plus gel or to Monovisc

Inclusion Criteria: patients with Osteoarthritis grade II and III according to Kellgren and Lawrence grading were included.

Exclusion Criteria: patients with autoimmune illnesses, active inflammation or infected processes, anticoagulant, and known allergy to hyaluronic acid.

Target parameters:

* Lower extremity functional scale
* Visual analogue scale
* Range of motion
* Kellgren and Lawrence class grade

Eligibility:

Ages Eligible for Study: 20 years to 70 years Genders Eligible for Study: both Accepts Healthy Volunteers: no

Criteria

Inclusion Criteria:

* Age of patients between 20 and 70 years
* patients with Osteoarthritis grade II and III according to Kellgren and Lawrence grading

Exclusion Criteria:

* Autoimmune illnesses
* Active inflammation or infected processes
* Anticoagulant
* Known allergy to hyaluronic acid.

ELIGIBILITY:
Inclusion Criteria:

* Age of patients between 20 and 70 years
* patients with Osteoarthritis grade II and III according to Kellgren and Lawrence grading

Exclusion Criteria:

* Autoimmune illnesses
* Active inflammation or infected processes
* Anticoagulant
* Known allergy to hyaluronic acid.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient with knee osteoarthiritis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Lower extremity functional scale | up to 52 weeks

SECONDARY OUTCOMES:
Visual analog scale | up to 52 weeks
Kellgren and lawrence class grade | up to 52 weeks
Range of motion | up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Hafez, Professor, Principal Investigator — October 6 University; Abdullah I Ammoura, Researcher, Study Chair — Bone and Joint Center
Locations (1):
- October 6 University, Six October City, Egypt